CLINICAL TRIAL: NCT02916576
Title: User Performance Evaluation of Contour® Plus One, Accu-Chek® Performa Connect, FreeStyle Optium Neo and OneTouch® Select Plus Blood Glucose Monitoring Systems Following ISO 15197:2013; EN ISO 15197:2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: IDT-1616-AL
Record Dates: First submitted 2016-09-06; First posted 2016-09-27 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Self-Testing

ARMS (1):
- Blood glucose measurement (Experimental)
  Interventions: Device: Blood-Glucose Monitoring Systems for self-testing

INTERVENTIONS:
Device: Blood-Glucose Monitoring Systems for self-testing — This is a user performance study, that is intended to show whether people with diabetes are able to obtain accurate measurement results with a blood glucose monitoring system (BGMS).
  The subjects' measurement technique (e.g. applying blood onto the system reagent, reading the result) will be observed and documented by study personnel.
  Immediately after the measurement by the subject, the study personnel will perform a measurement with the same test meter.
  Measurement results obtained by the subjects with the BGMS will be compared to measurement results obtained with the comparison method.
  Sample collection for the comparison measurement will be performed by study personnel within 5 min after the subject's measurement with the test meter.
  The samples will be collected from the subjects' skin puncture (if possible), an additional skin puncture (if required) will be documented.
  An additional skin puncture will be performed by study personnel with single-use lancing devices.
  Other Names: Contour Plus One, Accu-Chek Performa Connect, FreeStyle Optium Neo and OneTouch Select Plus

SUMMARY:
The user performance evaluation shows whether people with diabetes are able to obtain accurate measurement results with a blood glucose monitoring system. In this study, user performance evaluation will be performed for Contour Plus One (Ascensia Diabetes Care GmbH), Accu-Chek Performa Connect (Roche Diabetes Care GmbH), FreeStyle Optium Neo (Abbott Diabetes Care Inc.), OneTouch Select Plus (LifeScan Europe) based on ISO 15197:2013; EN ISO 15197:2015, clause 8.

For each BGMS, measurement procedures for user performance evaluation will be performed with 1 test meter and 1 reagent system lot by the study subjects.

The same meter and an additional test meter will be used for double measurements performed by study personnel (with the same reagent system lot used by subjects).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with type 1 diabetes, type 2 diabetes or subjects without diabetes
* Signed informed consent form
* Minimum age of 18 years
* Subjects are legally competent and capable to understand character, meaning and consequences of the study.
* If blood glucose values < 80 mg/dl or > 300 mg/dl shall be measured after short term alteration in insulin therapy:
* Male or female with type 1 diabetes and intensified insulin therapy or insulin pump therapy.
* Signature of subjects to document consent with these procedures on informed consent form.

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with potential risk during the test procedures (at the study physician's discretion)
* Current constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* Being unable to give informed consent
* < 18 years
* Legally incompetent
* Being committed to an institution (e.g. psychiatric clinic)
* Language barriers potentially compromising an adequate compliance with study procedures
* Dependent on investigator or sponsor
* If blood glucose values < 80 mg/dl shall be measured after short term alteration in insulin therapy, subjects with type 1 diabetes, suffering from:
* Coronary heart disease
* Condition after myocardial infarction
* Condition after cerebral events
* Peripheral arterial occlusive disease
* Hypoglycemia unawareness

Inclusion and exclusion criteria defined by ISO 15197:2013; EN ISO 15197:2015:

* Only subjects with diabetes type 1 or type 2 will be included.
* Demographic data will be collected to demonstrate that subjects represent different ages, genders and education levels.
* In deviation from ISO 15197:2013; EN ISO 15197:2015, included subjects may have participated in a study involving the BGMS, but must not yet have performed measurements with the BGMS according to their own statement for the last 3 years.
* In addtition, included subjects did not use the BGMS being evaluated at home for the last 3 years according to their own statement.
* In order to ensure that capillary blood samples meet the requirements indicated in the manufacturer's labelling,
* a physician will review the subjects' anamnesis and medication and check for interfering substances indicated in the manufacturer's labelling.
* the hematocrit value of each subject will be checked to be within the range indicated in the manufacturer's labelling (hematocrit determination before or after the measurement procedure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
System accuracy criteria (see description) | For each subject, the experimental phase has an expected duration of up to 3 hours
  Acceptance criteria defined by ISO 15197:2013 (E) / EN ISO 15197:2015 will be applied:
  95 % of the individual glucose measured values shall fall within ± 15 mg/dl (0.83 mmol/l) of the measured values of the comparison measurement procedure at glucose concentrations < 100 mg/dl (5.55 mmol/l) and within ± 15 % at glucose concentrations ≥ 100 mg/dl (5.55 mmol/l).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany

REFERENCES:
- [Derived] Freckmann G, Jendrike N, Baumstark A, Pleus S, Liebing C, Haug C. User Performance Evaluation of Four Blood Glucose Monitoring Systems Applying ISO 15197:2013 Accuracy Criteria and Calculation of Insulin Dosing Errors. Diabetes Ther. 2018 Apr;9(2):683-697. doi: 10.1007/s13300-018-0392-6. Epub 2018 Mar 3. PMID 29502304